CLINICAL TRIAL: NCT06094426
Title: A Single-arm Clinical Study of Autologous Tumor-infiltrating Lymphocyte Injections for the Treatment of Advanced Solid Tumors
Brief Title: Autologous Tumor Infiltrating Lymphocyte Injection for the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-316-001
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor; Adult; GT316

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GT316 treatment group (Experimental)
  Interventions: Biological: GT316

INTERVENTIONS:
Biological: GT316 — Autologous Tumor Infiltrating Lymphocyte Injection

SUMMARY:
This trial is a multicenter, single-arm, open design designed to evaluate the safety and tolerability of Autologous Tumor Infiltrating Lymphocyte Injection in the treatment of patients with advanced solid tumors, as well as pharmacokinetic profiling and efficacy. The trial consists of two phases: dose-escalation and dose-expansion.

ELIGIBILITY:
Inclusion Criteria:

* 1.The Patients (or legally authorized representative) Patients (or legally authorized representative) must have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC), must have the ability to understand the requirements of the study;
* 2.Must have a confirmed diagnosis of malignancy of their receptive histologies or cytologies: unresectable recurrent or metastatic solid tumor;
* 3.At least one resectable lesion (preferably superficial metastatic lymph nodes) that has not been treated with radiation and has not received other local therapies. The separated tissues ≥1.0cm^3 (either of single lesion origin or multiple lesions combined) for the preparation of autologous tumor-infiltrating lymphocytes. Minimally invasive treatment where possible;

Exclusion Criteria:

* 1.Patients with ≥3 untreated CNS metastases at the time of screening (patients were included if they had ≤3 CNS metastases with a maximum diameter of <1 cm and no peritumor edema on brain imaging (MRI or CT) and no evidence of progressive CNS disease on brain imaging for at least 3 months after treatment)
* 2.The patient who has any active autoimmune disease, history of autoimmune disease, need for systemic steroid hormones or a condition requiring immunosuppressive drug therapy (>10 mg/day of prednisone or equivalent hormone);
* 3. Arterial/venous thrombotic events within 3 months prior to enrollment, such as: cerebrovascular accident, deep vein thrombosis and pulmonary embolism occurring;
* 4.Patients with refractory or intractable epilepsy, drug-uncontrolled pleural effusion, abdominal effusion, pericardial effusion, active gastrointestinal bleeding or contraindications to IL-2;
* 5. Participate in other clinical trials within 4 weeks prior to screening, or planning to participate in this study and other clinical trials at the same；
* 6. Patients who have received allogeneic bone marrow transplantation or an organ allograft;
* 7.Patients who have a history of hypersensitivity to any component or excipient of study drugs: autologous tumor infiltrating lymphocytes, cyclophosphamide, fludarabine, IL-2, dimethyl sulfoxide (DMSO), human serum albumin (HSA), dextran-40 and antibiotics (beta lactam antibiotics, gentamicin);

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-26 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events per CTCAE 5.0 | 3 years
  To characterize the safety profile of autologous TIL injection in patients with relapsed/metastatic advanced solid tumor as measured by the incidence and severity of adverse events per CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No